CLINICAL TRIAL: NCT00069745
Title: A Multi-National Phase III Study of Satraplatin Plus Prednisone or Placebo Plus Prednisone in Patients With Hormone Refractory Prostate Cancer Previously Treated With One Cytotoxic Chemotherapy Regimen
Brief Title: Satraplatin in Hormone Refractory Prostate Cancer Patients Previously Treated With One Cytotoxic Chemotherapy Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPC SAT3-03-01
Record Dates: First submitted 2003-09-30; First posted 2003-10-06 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer; Hormone Refractory Prostate Cancer
Keywords: Prostatic Neoplasms; Cancer Treatment Protocols; Antineoplastic protocols; One Prior Cytotoxic Chemotherapy Regimen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — satraplatin; Prednisone

INTERVENTIONS:
Drug: Satraplatin
Drug: Prednisone

SUMMARY:
PURPOSE:

The SPARC trial is designed to compare the combination of the investigational oral cytotoxic drug, satraplatin, and prednisone, versus prednisone alone as second line chemotherapy in patients with hormone-refractory prostate cancer (HRPC).

TARGET PATIENT POPULATION:

The SPARC trial is intended for patients who have hormone-refractory prostate cancer (HRPC) and whose disease has progressed after treatment with one chemotherapy regimen. Please refer to the Eligibility Criteria page for the key inclusion and exclusion criteria.

WHAT IS SATRAPLATIN:

Satraplatin is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally. Satraplatin is also the only platinum-based drug that has demonstrated efficacy against prostate cancer in a randomized trial.

RATIONALE:

There are currently no approved chemotherapy drugs for the second line treatment of hormone-refractory prostate cancer (HRPC). In a preliminary randomized trial conducted in Europe, the combination of satraplatin and prednisone had superior activity compared to prednisone alone, for the treatment of HRPC patients who had not previously been treated with chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Stage D2 metastatic prostate cancer
* Progression after one prior chemotherapy
* ECOG Performance status equal / less than 2
* Life expectancy > 3 months
* Surgical or medical castration
* Adequate bone marrow, hepatic and renal functions
* Informed consent

Exclusion Criteria:

* More than one prior chemotherapy
* Prior platinum containing compounds
* Prior malignancy
* Prior significant RT/radionuclide therapy
* Major GI surgery or GI disease affecting absorption
* Disease with contraindication to steroids
* Brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Primary Completion 2006-01 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (210):
- United States (104):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology & Oncology Assoc., Sedona, Arizona
  - Hematology Oncology Physicians/SMO, Tucson, Arizona
  - Arizona Cancer Center, Tuscon, Arizona
  - California Cancer Center, Fresno, California
  - Pacific Shores Medical Group, Long Beach, California
  - Division of Hematology - Oncology, Los Angeles, California
  - University of California Davis Cancer Center, Division of Hematology-Oncology, Sacramento, California
  - Sharp Healthcare - Clinical Oncology Research, San Diego, California
  - Rocky Mountain Cancer Center - Midtown, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - DeQuattro Community Cancer Center, Manchester, Connecticut
  - Cancer Centers of Florida-Altamonte, Altamonte Springs, Florida
  - The Center for Hematology Oncology, Boca Raton, Florida
  - Hematology/Oncology Group of South Florida, Miami, Florida
  - Innovative Medical Research of South Florida, Miami Shores, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - South Florida Oncology & Hematology, Plantation, Florida
  - Hematology/Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Oncology and Hematology Associates of West Broward P.A., Tamarac, Florida
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwest Medical Specialists, Niles, Illinois
  - North Shore Research Association, Skokie, Illinois
  - Central Indiana Cancer Centers, Fishers, Indiana
  - Indiana Hematology Oncology Consultants, Indianapolis, Indiana
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Oncology Associates of Cedar Rapids, Cedar Rapids, Iowa
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - LSU Health Science Center, Stanley S. Scott Cancer Center, New Orleans, Louisiana
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - Berkshire Hematology Oncology, Pittsfield, Massachusetts
  - Karmanos Cancer Institute, Wayne State University, Detroit, Michigan
  - Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Hematology/Oncology Consultants, Inc., St Louis, Missouri
  - Arch Medical Services, Inc., Washington, Missouri
  - Nebraska Methodist Hospital Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology PA, Hooksett, New Hampshire
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Lovelace Sandia Health Systems, Albuquerque, New Mexico
  - Veterans Affairs Medical Center, Albuquerque, New Mexico
  - The University of New Mexico, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Albany Regional Cancer Center, Albany, New York
  - New York Oncology Hematology, P.C., Albany, New York
  - Advanced Oncology Associates, Armonk, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Interlakes Oncology Hematology, Canandaigua, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - New York Oncology Hematology, Rexford, New York
  - VA Medical Center Syracuse, Syracuse, New York
  - Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - Piedmont Hematology - Oncology, Winston-Salem, North Carolina
  - Dayton Oncology Hematology, Kettering, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Hematology and Oncology Associates of Northeastern PA / PC, Dunmore, Pennsylvania
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Charleston Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Cancer Center of the Carolinas, Seneca, Seneca, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Texas Cancer Center, Abilene, Texas
  - Texas Oncology, Arlington, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Onoclogy PA - Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - The Texas Cancer Center, Dallas, Texas
  - TOPA Sammons Cancer Center, Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - San Antonio Tumor & Blood Clinic, Fredericksburg, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Texas Oncology, P.A. - Irving, Irving, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - S. Texas Cancer Center, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Allison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Hematology Oncology Associates of South Texas, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Waco Cancer Care Research Center, Waco, Texas
  - Texas Oncology, P.A. - Deke Slayton Cancer Center, Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc., Salem, Virginia
  - Puget Sound Cancer Center - Edmonds, Edmonds, Washington
  - Cancer Care Northwest-North, Spokane, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Argentina (16):
  - Hospital Italiano de Buenos Aires, Capital Federal, Buenos Aires
  - Clinica Oncologica de Excelencia, Capital Federal, Buenos Aires
  - Policlinica Bancaria "9 de Julio" Av. Gaona 2197, Capital Federal, Buenos Aires
  - Hospital General de Agudos E. Tornu, Capital Federal, Buenos Aires
  - Salisbury Investigaciones Clinicas del Grupo CER S.A., Quilmes, Buenos Aires
  - Hospital Italiano Regional del Sur Dept. Oncology, Bahía Blanca
  - Grupo Plaza Dept. Oncology, Belén de Escobar
  - Instituto Quirúrgico del Callao, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Centro Oncológico LALCEC, Concepcion Del Uruguay, Entre Ríos
  - Hospital Italiano de Cordoba Dept. Oncology, Córdoba
  - Unidad Oncologica del Neuquen, Neuquén
  - Caici Dept. Oncology, Rosario
  - Centro Oncologico Rosario, Rosario
  - Centro San Roque, San Miguel de Tucumán, Tucumán
  - Clinical Especializada ISIS, Santa Fe
- Belgium (5):
  - AZ-VUB, Brussels
  - Institut Jules Bordet Service de Chimiothérapie, Brussels
  - Hopital Erasme, Brussels
  - UCLC St. Luc, Brussels
  - Sint Maartenziekenhuis, Kortrijk
- Croatia (2):
  - Clinical Hospital Split Department of Oncology and Radiotherapy, Split
  - Clinical Hostpital Rebro Department of Oncology, Zagreb
- France (17):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Hôpital de La Tronche - CHU de Grenoble: Departement de cacerologie et d'hematologie, Grenoble
  - Clinique du Mail Service d'Oncologie, Grenoble
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - Chu Dupuytren, Limoges
  - CRLC Léon Bérard, Lyon
  - Centre Hospitalier Belfort-Montbeliard, Montbéliard
  - CRLC Val d'Aurelle Paul-Lamarque, Montpellier
  - Centre Antoine Lacassagne Oncologie medicale, Nice
  - Hôpital Saint-Louis: Service de Radiotherapy, Paris
  - Hôpital Tenon, Paris
  - CHU de Poitiers, Poitiers
  - Institut Jean , Service d'Oncologie, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (18):
  - RWTH Aachen, Aachen
  - Vivantes Krankenhaus am Urban, Berlin
  - Fach- und Belegarzte fur Urologie, Berlin
  - Diakonissenkrankenhaus Dessau gGmbH, Dessau
  - Universitätsklinikum der Carl-Gustav-Carus Universität, Dresden
  - Stadtische Klinicen Frankfurt a.M. Hochst, Frankfurt a.M. Hochst
  - EuromedClinic, Fürth
  - Klinikum der medizinischen Fakultät der Martin-Luther-Universität Halle-Wittenberg, Halle
  - Niedergelassener Urologe, Hamburg
  - Medizinische Hochschule, Hanover
  - Marienhospital II, Herne
  - Universitatklinikum Schleswig-Holstein, Lübeck
  - Klinickum der Johannes-Gutenberg Universitat, Mainz
  - Klinikum der Philipps - Universitat Marburg, Marburg
  - Klinikum rechts der Isar, München
  - Universitatklinikum Munster, Münster
  - Klinik Bad Trissel, Oberaudorf
  - Urologische Praxis, Saarbrücken
- Hungary (4):
  - St. Margit Hospital, Budapest
  - St. Istvan Hospital, Budapest
  - National Institute of Oncology, Budapest
  - Pecs Medical University, Pécs
- Israel (4):
  - Soroka Medical Center, Beerhseva
  - Rambam Medical Center, Haifa
  - Hadassah University, Jerusalem
  - Hospital Ein Kerem Asaf Harofeh Medical Center, Ẕerifin
- Italy (6):
  - Istituto Nazionale per la Ricerca sul Cancro (IST), Genoa
  - Universita degli Studi di Napoli Federico II-Nuovo Policlinico, Napoli
  - A.S.O. San Luigi, Orbassano
  - Azienda Ospedaliera di Padova, Padua
  - A.O. San Camillo-Forlanini, Rome
  - Istituto Clinico Humanitas: Dipartimento di Oncologia Medica ed Ematologia, Rozanno (MI)
- Netherlands (3):
  - Academic Hospital of the University of Amsterdam, Amsterdam
  - Academisch Ziekenhuis Nijmegen: Urology Department, Nijmegen
  - Streekziekenhuis Koningin : Dept. Urology, Winterswijk
- Peru (3):
  - Essalud Dept. Oncology, Jesus Maria
  - San Felipe (Oncomedical), Lima
  - INEN Dept Onco-Hemato, Lima
- Poland (8):
  - Oddzial Chemioterapii, Bialostocki Osrodek Onkologiczny, Bialystok
  - Oddzial Onkologii I Radioterapii, Szpital Morski im. PCK, Gdynia
  - Akademia Medyczna w Lodzi, Lodz
  - Akademia Medyczna w Lublinie, Lublin
  - Oddzial Radioterapii, Wielkopolskie Centrum Onkologii - Instytut, Poznan
  - Akademia Medyczna w Szczecinie, Szczecin
  - Klinika Nowotworow Ukladu Moczowego, Centrum Onkologii - Instytut, Warsaw
  - Oddzial Chemioterapii, 4 Wojskowy Szpital Kliniczny, Wroclaw
- Russia (3):
  - N.N Blokchin Cancer Research Centre, Moscow
  - Hertzen Research Institute of Oncology, Moscow
  - Medical Radilogical Research Center of Rams, Obninsk
- Spain (7):
  - Hospital de la Santa Creu i Sant Pau, Sevicio de Oncología Médica, Barcelona
  - Hospital Clinic i Provincial, Sevicio de Oncología Médica, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clínico San Carlos, Sevicio de Oncología Médica, Madrid
  - Clinica Universitaria de Navarra, Sevicio de Oncología Médica, Pamplona
  - Hospital Universitario Marqués de Valdecilla, Sevicio de Oncología Médica, Santander
  - Instituto Valenciano de Oncología: Sevicio de Oncología Médica, Valencia
- United Kingdom (10):
  - Aberdeen Royal Infirmary, Aberdeen
  - CRUK Institute for Cancer Studies, Birmingham
  - Bristol Oncology Centre, Bristol
  - Beatson Oncology Center, Glasgow
  - Guy's hospital, London
  - St George's Healthcare Dept of Oncology, Tooting, London
  - St. Bartholomew's Hospital Dept. of Medical Oncology, London
  - Northern Centre for Cancer Treatment, Newcastle upon Tyne
  - Lister Hospital Department of Urology, Stevenage Hertfordshire
  - Royal Marsden Hospital, Sutton